CLINICAL TRIAL: NCT02360436
Title: EPITRA-14-001: Analysis of the Glutathione Cycle in Children With Rett Syndrome
Brief Title: Analysis of the Glutathione Cycle in Children With Rett Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Priorities other studies
Sponsor: Edison Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EPITRA-14-001
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Rett Syndrome
Keywords: Rett; MeCP2; Glutathione; Cysteine; ROS
MeSH Terms: conditions — Rett Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Analyis of the Glutathione Cycle in Children with Rett Syndrome

DETAILED DESCRIPTION:
To analyze the levels of glutathione and relevant glutathione metabolites in children with Rett syndrome in an effort to better understand disease pathology and biochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Age between 2 and 10, inclusive
* Genetically-confirmed diagnosis of Rett syndrome with MeCP2 mutation
* No change in dietary supplements in three months prior to the initial blood draw
* No participation in interventional pharmaceutical clinical trials in prior 12 months

Exclusion Criteria:

* None other than meeting Inclusion criteria

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-10 with genetically confirmed diagnosis of Rett syndrome with MeCP2 mutation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2015-07-31 (Estimated); Study Completion 2015-09-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of changes in levels of glutathione and relevant glutathione metabolites in children with Rett syndrome from baseline to the end of month 6 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alan Percy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States